CLINICAL TRIAL: NCT01849224
Title: Randomized Trial of Pelvic and Lower Extremity Exercise in Patients Who Underwent Pelvic Lymphadenectomy With Lower Extremity Edema-related Symptoms
Brief Title: Randomized Trial of Exercise on Lower Extremity Edema After Lymphadenectomy in Gynecologic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Myong Cheol Lim, Senior researcher, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCNCS-13-723
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Gynecologic Cancer
Keywords: Lower extremity edema; Lower leg lymphedema; Lower leg edema; Lymphedema; Pelvic lymphadenectomy; Exercise
MeSH Terms: conditions — Lymphedema; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pelvic and lower extremity exercise (Experimental): Experimental arm will be educated the guidelines for prevention and early detection of lower extremity edema. Additionally, pelvic and lower extremity exercise will be educated and participants will continue exercise for 1 year at home.
  Interventions: Other: Pelvic and lower extremity exercise
- Control (No Intervention): Control group will be educated the guidelines for prevention and early detection of lower extremity edema

INTERVENTIONS:
Other: Pelvic and lower extremity exercise
  Arms: Pelvic and lower extremity exercise

SUMMARY:
The primary outcome is the change in lower extremity edema-related symptoms. Secondary outcomes include the compliance rate of management guidelines for lower extremity edema, the performance rate for pelvic and lower extremity exercise.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age
* Patients who underwent pelvic lymphadenectomy
* Patients with suspicious pelvic cancer who finished active treatments such as chemotherapy, radiotherapy or surgery. The interval between the time of randomization and the end of the treatment should be more than 2 weeks.
* The patient is able to understand the study and is willing to give written informed consent to the study
* patient with edema-related symptoms such as leg heaviness, distension, tightness, pain, limited movement, or weakness etc.

Exclusion Criteria:

* Severe systemic diseases causing peripheral edema, including renal disease
* Severe or uncontrolled cardiopulmonary disease, including implantable device such as a pacemaker
* Acute superficial or deep vein thrombosis
* Previous major surgery for lower extremities, including metallic surgical implant
* Local infection in the lower extremities
* Auto-immunological disorders or vasculitis
* Use of systemic corticosteroids
* Pregnant or currently breastfeeding
* Alcohol or drug abuse
* Uncontrolled diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in lower extremity edema-related symptoms after pelvic and lower extremities exercise | 1 year after randomization

SECONDARY OUTCOMES:
the compliance rate of management guidelines for lower extremity edema, the performance rate for pelvic and lower extremity exercise | 1 year after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Lim Myong Cheol, MD,PhD, Principal Investigator — National Cancer Center
Locations (1):
- Myong Cheol Lim, Goyang-si, Gyeonggi-do, South Korea